CLINICAL TRIAL: NCT02268435
Title: A Trial of Dovitinib in Combination With Imatinib in Patients With Metastatic or Unresectable Gastrointestinal Stromal Tumors After Failure to Imatinib and Sunitinib
Brief Title: Dovitinib in Combination With Imatinib in Patients With Gastrointestinal Stromal Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Dovitinib Production stopped
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1401
Record Dates: First submitted 2014-10-07; First posted 2014-10-20 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dovitinib plus Imatinib (Experimental): Dovitinib once daily on a 5 days on/2 days off dosing schedule, and imatinib once daily on a continuous dosing schedule
  Interventions: Drug: dovitinib plus imatinib

INTERVENTIONS:
Drug: dovitinib plus imatinib — Dovitinib once daily on a 5 days on/2 days off dosing schedule, and imatinib once daily on a continuous dosing schedule

SUMMARY:
The objective of this study is to determine the recommended dose of combination of dovitinib and imatinib in phase I study.

DETAILED DESCRIPTION:
combination of dovitinib and imatinib could lead to additive or synergistic effect in patients who had failure of standard TKI therapies including imatinib, sunitinib, and/or regorafenib. In this phase I-II study of dovitinib plus imatinib, we aim to determine a recommended dose of dovitinib plus imatinib and to evaluate the safety and activity of the combination at the recommended dose as a 3rd or more line of treatment in metastatic or unresectable GIST.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 years or older
2. Histologically confirmed metastatic or unresectable GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRα gene
3. Disease control (response or stabilization for at least 6 months with first-line imatinib and failure of prior treatments for GIST, including at least both imatinib and sunitinib and/or regorafenib. However, patients with imatinib rechallenge will not be accrued.
4. ECOG performance status of 0~2
5. Resolution of all toxic effects of prior treatments to grade 0 or 1
6. At least one evaluable or measurable lesion for phase I study
7. Adequate bone marrow, hepatic, renal, and other organ functions

   * Neutrophil > 1,500/mm3
   * Platelet > 75,000/mm3
   * Hemoglobin > 8.0 g/dL
   * Total bilirubin < 1.5 x upper limit of normal
   * AST/ALT < 2.5 x ULN with no exceptions
   * Creatinine < 1.5 x ULN
8. Life expectancy > 12 weeks
9. Women with reproductive potential must have a negative serum or urine pregnancy test; and men and women of reproductive potential must practice an effective method of avoiding pregnancy while receiving study drug.
10. Washout period of previous TKIs or chemotherapy for more than 4 times the half life.
11. No prior use of dovitinib or other inhibitors of FGFR except regorafenib
12. Provision of a signed written informed consent

Exclusion Criteria:

1. Women of child-bearing potential who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial in both sexes.
2. Clinically significant cardiac disease or impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * LVEF < 45%
   * Complete left bundle branch block
   * Obligate use of a cardiac pacemaker
   * Congenital long QT syndrome
   * History or presence of ventricular tachyarrhythmia
   * Presence of unstable atrial fibrillation .
   * Clinically significant resting bradycardia
   * Uncontrolled hypertension
   * QTc > 480 msec on screening ECG
   * Right bundle branch block + left anterior hemiblock
   * Angina pectoris ≤ 3 months prior to starting study drug
   * Acute Myocardial Infarction ≤ 3 months prior to starting study drug
   * Other clinically significant heart disease
3. Uncontrolled infection
4. Subjects who did not tolerate previous imatinib treatment.
5. Diabetes mellitus with signs of clinically significant peripheral vascular disease
6. Previous pericarditis; clinically significant pleural effusion in the previous 12 months or current ascites requiring two or more interventions/month 7. Known pre-existing clinically significant disorder of the hypothalamic-pituitary axis, adrenal or thyroid glands

8. Prior acute or chronic pancreatitis of any etiology 9. Malabsorption syndrome or uncontrolled gastrointestinal toxicities with toxicity greater than NCI CTCAE grade 2 10. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for this study 11. Treatment with any of the medications that have a potential risk of prolonging the QT interval or inducing Torsades de Points and the treatment cannot be discontinued or switched to a different medication prior to starting study drug 12. Use of ketoconazole, erythromycin, carbamazepine, phenobarbital, rifampin, phenytoin and quinidine 2 weeks prior baseline 13. Major surgery ≤ 28 days prior to starting study drug or who have not recovered from side effects of such therapy 14. Known diagnosis of HIV infection 15. History of another primary malignancy that is currently clinically significant or currently requires active intervention 16. Patients with brain metastases as assessed by radiologic imaging due to symptoms clinically suspected of brain metastases 17. Alcohol or substance abuse disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose and recommended dose | 3 years
  Initially three patients will be treated at each dose level. If one out of three patients experiences a DLT, three additional patients will be entered at that dose level. Dose escalation will be continued until DLTs are experienced in two or more out of six patients (more than 33% of patient cohort), which will be defined as the MTD.If more than 33% of patients experience a DLT in a dose level, one doe level below will be the RD

SECONDARY OUTCOMES:
Disease control rate | 3 years
  response + stable disease evaluated with abdominal and pelvic spiral CT scan every 4 weeks for the first 8 weeks, and then every 8 weeks, using RECIST criteria v1.1
Overall response rate | 3 years
  response + stable disease evaluated with abdominal and pelvic spiral CT scan every 4 weeks for the first 8 weeks, and then every 8 weeks, using RECIST criteria v1.1
Number of Participants with Adverse Events as a Measure of Safety | 3 years
  Safety by NCI CTCAE version 4.0
Progression-free survival | 3 years
  response + stable disease evaluated with abdominal and pelvic spiral CT scan every 4 weeks for the first 8 weeks, and then every 8 weeks, using RECIST criteria v1.1
Overall survival (OS) | 3 years
  OS assessment dates will be the time point when 6 months have passed after the enrollment of the last patient
optionally, correlation of efficacy with potential biomarkers | 3 years
  mutational analysis of KIT exons 9, 11, 13, and 17, and PDGFRα exons 12, 14, and 18 with direct sequencing using DNA extracted from archival tissues and/or newly obtained tissues at baseline, and with BEAMing assay using ctDNA extracted from plasma at baseline and every time when follow-up CT scans are conducted; optionally circulating growth factors including but not limited to VEGF, bFGF, IL-8, PLGF, FGFR2, and FGF23, and soluble receptors including but not limited to sVEGFR1 and 2 with plasma collected at baseline and on Cycle 1 Week 4 Day 5
next generation sequencing will be performed in newly obtained tissues at baseline to find out new genetic changes after failure of previous standard TKIs | 3 years
Optionally, activation of FGFR signaling will be analyzed using the reverse phase protein microarray and/or immunohistochemistry including but not limited to pFRS2 and pFGFR in archival tissues and/or newly obtained tissues at baseline | 3 years
Imatinib and dovitinib plasma concentrations vs time profile, and basic pharmacokinetics parameters | 3 years
  PK samples will be taken at 0 hour (pre-dose) and at 1, 2, 3, 4, 6, and 8 hours (post-dose) after administration of dovitinib and imatinib on Cycle 1 Week 1 Day 1, Cycle 1 Week 1 Day 5, and Cycle 1 Week 4 Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, PhD, Principal Investigator — Asan Medical Center